CLINICAL TRIAL: NCT01265524
Title: A Phase 2, Randomized, Double-Blind, Multi-center Study Comparing CLP Versus Placebo in Heart Failure Patients With Chronic Kidney Disease
Brief Title: Evaluation of CLP in Heart Failure Patients With Chronic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sorbent Therapeutics (Industry)
Collaborators: Pharmaterra (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CTST-21
Record Dates: First submitted 2010-12-20; First posted 2010-12-23 (Estimated); Results first posted 2013-03-13 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CLP (Active Comparator): Investigational drug: 15 g CLP per day given as capsules
  Interventions: Drug: CLP
- Placebo (Placebo Comparator): Placebo, capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CLP — Oral administration
  Arms: CLP
Drug: Placebo — Oral administration
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effects of CLP on serum potassium and signs and symptoms of fluid overload in heart failure patients with chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure with New York Heart Association (NYHA) Classification III or IV
* Hospitalization for heart failure decompensation associated with fluid overload within the last six months
* Chronic kidney disease
* Must be able to understand study procedures and willing and able to provide written informed consent

Exclusion Criteria:

* No hospitalization within 4 weeks of Baseline Visit
* In the investigator's judgment, any cardiovascular, renal, hepatic, endocrine, gastrointestinal, neurological or other disease or condition that makes the patients study participation unsafe
* History or presence of gastrointestinal conditions such as severe constipation or gastrointestinal tract strictures
* Current dialysis patient, or anticipated need for dialysis during study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2011-04; Primary Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Detlef Albrecht, MD, Study Chair — Sorbent Therapeutics
Locations (3):
- Yerevan, Armenia
- Tbilisi, Georgia
- Chisinau, Moldova

REFERENCES:
- [Result] Costanzo MR, Heywood JT, Massie BM, Iwashita J, Henderson L, Mamatsashvili M, Sisakian H, Hayrapetyan H, Sager P, van Veldhuisen DJ, Albrecht D. A double-blind, randomized, parallel, placebo-controlled study examining the effect of cross-linked polyelectrolyte in heart failure patients with chronic kidney disease. Eur J Heart Fail. 2012 Aug;14(8):922-30. doi: 10.1093/eurjhf/hfs074. Epub 2012 May 21. PMID 22613585

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Although 113 subjects were randomized, 2 subjects did not receive study drug and were removed from the analysis as pre- specified in the SAP.
Groups:
- Investigational Drug: CLP: Investigational drug: 15 g CLP per day given as capsules
- Placebo: Placebo: capsules
Period: Overall Study
Arm/Group | Investigational Drug: CLP | Placebo
Started | 59 | 52
Completed | 41 | 46
Not Completed | 18 | 6

BASELINE CHARACTERISTICS:
Groups:
- Investigational Drug: CLP: Investigational drug: 15g CLP per day given as capsules
- Total: Total of all reporting groups
Arm/Group | Investigational Drug: CLP | Placebo | Total
Number analyzed (Participants) | 59 | 52 | 111
Age, Customized [Mean (Standard Deviation); unit: years] | 68 (8) | 70 (10) | 69 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 23 | 40
  Male | 42 | 29 | 71
Weight [Mean (Standard Deviation); unit: kg] | 75.3 (13.6) | 75.1 (16.2) | 75.2 (14.9)
eGFR [Mean (Standard Deviation); unit: ml/min/1.73m3] | 45.0 (14.2) | 44.9 (17.3) | 45 (15.8)
New York Heart Association (NYHA) Functional Class [Number; unit: participants] — NYHA Functional Classes are I, II, III, and IV A brief summary of the classes is included below. Class I: patients with cardiac disease but without resulting limitations of physical activity Class II: patients with cardiac disease with slight limitations to physical activity Class III: patients with cardiac disease with marked limitations of physical activity Class IV: patients with cardiac disease resulting in an inability to carry out physical activity without discomfort
  participants
    II | 0 | 2 | 2
    III | 52 | 45 | 97
    IV | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Potassium
Description: Change in serum potassium from baseline to Week 8.
Time Frame: Baseline and 8 weeks
Population: The efficacy and the safety analyses were done using the ITT population with Week 8/EOS data for the patients who did not complete the 8-week treatment period excluded. The ITT population included all randomized patients who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Investigational Drug: CLP | Placebo
Number analyzed (Participants) | 41 | 46
mg/dl | 0.15 (0.348) | 0.05 (0.345)

2. Secondary Outcome: Weight Loss at Week 1
Time Frame: Baseline and 1 week
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Investigational Drug: CLP | Placebo
Number analyzed (Participants) | 56 | 52
kg | -0.71 (1.5) | 0.11 (2.0)
Statistical Analysis 1: Comparison: Investigational Drug: CLP vs Placebo; Test type: Non-Inferiority or Equivalence — The efficacy and the safety analyses were done using the ITT population with Week 8/EOS data for the patients who did not complete the 8-week treatment period excluded. The ITT population included all randomized patients who received at least 1 dose of study drug; p = 0.014, ANCOVA — Corrections for multiplicity were not performed and P values < 0.05 were considered statistically significant; Continuous or ordinal data were analyzed using RM-ANCOVA using change from baseline values to compare CLP and placebo treatments

3. Secondary Outcome: Weight Loss at Week 2
Time Frame: Baseline and 2 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Investigational Drug: CLP | Placebo
Number analyzed (Participants) | 52 | 51
kg | -0.83 (1.8) | 0.29 (2.3)

4. Secondary Outcome: Frequency of Marked or Disabling Exertional Dyspnea by Physician Assessment at Week 4
Description: The frequency of marked or disabling exertional dyspnea was physician assessed based on physical exam at week 4.
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Investigational Drug: CLP | Placebo
Number analyzed (Participants) | 47 | 48
participants | 10 | 14

5. Secondary Outcome: Frequency of Marked or Disabling Exertional Dyspnea by Physician Assessment at Week 8
Description: The frequency of marked or disabling exertional dyspnea was physician assessed based on physical exam at week 8.
Time Frame: 8 weeks
Measure: Number; unit: participants
Arm/Group | Investigational Drug: CLP | Placebo
Number analyzed (Participants) | 41 | 46
participants | 5 | 12

6. Secondary Outcome: Number of Patients Improving by at Least One NYHA Functional Class From Baseline to Week 8
Time Frame: Baseline and 8 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Investigational Drug: CLP | Placebo
Number analyzed (Participants) | 41 | 46
participants | 20 | 8
Statistical Analysis 1: Comparison: Investigational Drug: CLP vs Placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.0002, ANCOVA — Corrections for multiplicity were not performed and P values < 0.05 were considered statistically significant; [statistical method as in outcome 2, analysis 1]

7. Secondary Outcome: 6MWT Distance at Week 8
Description: Increase in the 6 minute walk test (6MWT) distance from baseline to Week 8. The test was performed according to the American Thoracic Society (ATS)Guidelines 2002.
Time Frame: Baseline and 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: m
Arm/Group | Investigational Drug: CLP | Placebo
Number analyzed (Participants) | 41 | 46
m | 39.3 (53.39) | 19.7 (39.17)
Statistical Analysis 1: Comparison: Investigational Drug: CLP vs Placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.072, ANCOVA — Corrections for multiplicity were not performed and P values < 0.05 were considered statistically significant; [statistical method as in outcome 2, analysis 1]

ADVERSE EVENTS:
Arm/Group | Investigational Drug: CLP | Placebo
Serious Adverse Events (participants affected / at risk) | 4/59 | 1/52
Other Adverse Events (participants affected / at risk) | 21/59 | 13/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Drug: CLP (N=59) | Placebo (N=52)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 1 (1)
Sudden death (Cardiac disorders) | 1 (1) | 0 (0)
Renal failure (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Investigational Drug: CLP (N=59) | Placebo (N=52)
Abdominal discomfort (Gastrointestinal disorders) | 7 | 2
Abdominal distention (Gastrointestinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3
Oedema peripheral (General disorders) | 4 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypertension (Vascular disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A standard confidentiality agreement is in place.